CLINICAL TRIAL: NCT02918474
Title: Decision Making Tool for Contralateral Prophylactic Mastectomy
Brief Title: Decision Making Tool in Supporting Decision Making in Contralateral Prophylactic Mastectomy in Patients With Newly Diagnosed Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PA16-0469; NCI-2018-02660 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA16-0469 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Ductal Breast Carcinoma In Situ; Invasive Breast Carcinoma; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Sporadic Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (decision making tool) (Experimental): Patients use decision making tool during consultation with breast cancer surgeon and complete questionnaires before and after consultation.
  Interventions: Other: Decision Aid; Other: Questionnaire Administration

INTERVENTIONS:
Other: Decision Aid — Use decision making tool
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies the acceptability and how well decision making tool works in supporting decision making in contralateral prophylactic mastectomy in patients with newly diagnosed breast cancer. Decision making tool may help patients with early stage breast cancer make decisions regarding their surgical options.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. An online decision support tool will be field tested that provides patients facing a decision about contralateral prophylactic breast cancer (CPM) with evidence-based information about the expected incidence of contralateral breast cancer and the life expectancy benefit of CPM. The tool will be designed for use in clinical settings and viewed jointly by the patient and physician as part of a shared decision making process around CPM.

OUTLINE:

Patients use decision making tool during consultation with breast cancer surgeon and complete questionnaires before and after consultation.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed ductal breast carcinoma in situ (DCIS) or stage I-III sporadic unilateral invasive breast cancer
* Able to speak read or write English

Exclusion Criteria:

* Patients with previous breast cancer
* Prior history of bilateral prophylactic mastectomy
* Known to have a germline mutation that predisposes them to an increased risk of breast cancer (e.g. BRCA1/2) and/or they are considered at high risk for contralateral breast cancer on the basis of a strong family history of cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-04-28 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the decision support tool | Up to 2 years
  Patients' rating of the acceptability of the decision support tool will be assessed using questions from the Ottawa Acceptability Measures, including the clarity, amount, and balance of the information provided by the tool. Acceptability data from patients enrolled in the field test will be reported descriptively.
Changes in patient's knowledge of contralateral prophylactic mastectomy (CPM) | Baseline up to 2 years
  Will test for change in knowledge from before to after administration of the decision support tool with a breast cancer surgeon using paired samples t-tests.
Reductions in decisional conflict about CPM | Baseline up to 2 years
  Will be assessed using the Decisional Conflict Scale. Will test for reduction in decisional conflict from before to after administration of the decision support tool with a breast cancer surgeon using paired samples t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Abenaa M Brewster, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org